CLINICAL TRIAL: NCT03595995
Title: A Two-Stage, Randomized, Double-Blind, Dose-Ranging, Phase 2 Trial to Evaluate the Safety and Efficacy of UB-621 on HSV Shedding in Adults With Recurrent Genital HSV-2 Infection.
Brief Title: A Phase 2 Trial to Evaluate the Safety and Efficacy of UB-621
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: United BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UBP-A206-HSV
Record Dates: First submitted 2018-06-28; First posted 2018-07-23 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Genital Herpes
MeSH Terms: conditions — Herpes Genitalis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): 1. Placebo (volume equivalent to 2.5 mg/kg UB-621)
  2. 2.5 mg/kg UB-621
  Interventions: Biological: UB-621; Other: Placebo
- Cohort 2 (Experimental): 1. Placebo (volume equivalent to 5 mg/kg UB-621)
  2. 5 mg/kg UB-621
  Interventions: Biological: UB-621; Other: Placebo

INTERVENTIONS:
Biological: UB-621 — Monoclonal antibody by SC injection
Other: Placebo — The placebo is a sterile, clear and colorless or slightly yellow liquid, contains the same composition as UB-621 except drug substance. It is given by SC injection.

SUMMARY:
To evaluate the efficacy of two dose levels of UB-621 administration in reducing the HSV-2 genital shedding rate in patients with recurrent genital HSV-2 infection.

DETAILED DESCRIPTION:
This is a 2-stage, randomized, double-blind, dose-ranging, multi-center phase 2 study designed to evaluate the efficacy, safety, and PK of UB-621 given at 2.5 or 5 mg/kg in adult subjects with recurrent genital HSV-2 infection. The study consists of 2 stages of enrollments, in which 40 subjects will be enrolled in the first stage and randomly assigned to receive placebo or UB-621 at 2.5 mg/kg in a 1:3 ratio into Cohort 1 at Bv6 (Day B57), and another 40 subjects will be enrolled in the second stage and randomly assigned to receive placebo or UB-621 at 5 mg/kg in a 1:3 ratio into Cohort 2 at Bv6 (Day B57) after review by the Data Safety Monitoring Committee (DSMC). The DSMC will review safety data after all subjects of Cohort 1 complete the visit Fv6 (Day F28) and make the recommendation whether to proceed with enrollment for Cohort 2.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 18 years of age inclusive.
* Subject must be HSV-2 seropositive
* Subjects have a history of recurrent genital herpes in the past year
* Subjects have a negative result on the HIV Ab/Ag assay
* Subjects must agree to use contraception during study participation
* Subjects must be willing NOT to use any topical genital therapy and systemic anti-HSV therapy from the beginning of the study till the end of week 16.
* Subjects must be willing to collect a swab each day from their genital area (non-lesional as well as lesional, if appropriate) during the swabbing periods, which are 8 weeks prior to and upon the administration of study drug.
* Female subjects must have a negative serum β-HCG at Screening and a negative urine pregnancy test prior to study drug administration.

Exclusion Criteria:

* Serious medical conditions, including poorly controlled diabetes, significant autoimmune diseases, co-existing sexually transmitted disease presentation (except HSV) in the anogenital area, etc. that may interfere with the assessment of the efficacy of UB-621.
* Documented HSV resistance to acyclovir, valacyclovir, famciclovir, or penciclovir
* History or current evidence of malignancy except for a localized non-melanoma skin cancer
* Known immunosuppression
* Exposure to HSV vaccine
* Medical history of macular or maculopapular skin reactions to antibody (ie, as evidenced by IgG or plasma administration)
* Any other conditions that in the judgment of the Investigator would preclude successful completion of the clinical study
* Treatment with systemic steroids or other immunomodulating agents within 30 days prior to Screening or planned treatment with systemic steroids or immunomodulators during the study period.
* Renal impairment and/or hepatic impairment
* ECG abnormalities of clinical relevance or cardiovascular conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
change of HSV-2 shedding rate. | 112 days
  The primary endpoint for this study is to evaluate the reduction in HSV-2 shedding rate within subjects in the Baseline Period versus Follow-up Period.

SECONDARY OUTCOMES:
change of HSV-2 viral load | 112 days
  Anogenital swab samples collected from subjects during the Baseline Period and Follow-up Period will be used to quantify HSV-2 DNA copies to evaluate efficacy of UB-621 in reducing viral load.
change of genital lesion rates | 140 days
  Subject self-assessment of genital lesions will be recorded in subject diary as daily routine tasks from Bv1 (Day B1) until Fv11/EOS visit (Day F140). Data from subject self-assessment of genital lesions will be used to evaluate the efficacy of UB-621 in reducing genital lesions rates. Genital lesion rate will be measured by the number of days with lesion(s) reported divided by the number of days of study periods (Baseline Period, Transition Period, or Follow-up Period).
  Reduction in genital lesion rates will be evaluated before and after study drug treatment within subjects (Baseline versus Follow-up values).
Clinical and Subclinical HSV-2 Shedding Rates | 196 days
  Daily record of subject self-assessment of genital lesions in subject diary in addition to anogenital swabs collected daily from subjects during the Baseline and Follow-up Periods will be used to evaluate the efficacy of UB-621 in reducing clinical (lesional) and subclinical (non-lesional) HSV-2 shedding rates.
Rate of HSV-2 Shedding Episodes | 196
  Another secondary efficacy assessment includes the rate of HSV-2 shedding episodes as measured by the number of onsets of shedding episodes divided by the total number of days with swabs collected. Shedding episodes are defined as consecutive HSV-2 positive swab results including no more than 1 consecutive negative result or missed swab. The episodes are preceded and followed by 2 consecutive negative swab results.
  Daily record of subject self-assessment of genital lesions in subject diary in addition to anogenital swabs collected daily from subjects during the Baseline and Follow-up Periods will be used to evaluate the efficacy of UB-621 in reducing the rate of HSV-2 shedding episodes. Reduction in the rate of HSV-2 shedding episodes will be evaluated before and after study drug treatment within subjects (Baseline versus Follow-up values).